CLINICAL TRIAL: NCT00020527
Title: A Multicenter, Open, Non-Comparative, Sequential Dose-Escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Two Separate Doses of MK-0991 in Children With New Onset Fever and Neutropenia
Brief Title: Caspofungin Acetate in Treating Children With Fever and Neutropenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000068564; NCI-01-C-0084C; NCT00011219 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2003-03

CONDITIONS: Fever, Sweats, and Hot Flashes; Infection; Kidney Cancer; Leukemia; Lymphoma; Neuroblastoma; Neutropenia; Sarcoma
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood rhabdomyosarcoma; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; fever, sweats, and hot flashes; childhood acute promyelocytic leukemia (M3); recurrent/refractory childhood Hodgkin lymphoma; neutropenia; infection; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; previously treated childhood rhabdomyosarcoma
MeSH Terms: conditions — Fever; Hot Flashes; Infections; Kidney Neoplasms; Leukemia; Lymphoma; Neuroblastoma; Neutropenia; Sarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Wilms Tumor; Recurrence; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Caspofungin

INTERVENTIONS:
Drug: caspofungin acetate

SUMMARY:
RATIONALE: Giving caspofungin acetate may be effective in preventing or controlling fever and neutropenia caused by chemotherapy or bone marrow transplantation.

PURPOSE: Clinical trial to study the effectiveness of caspofungin acetate in treating children who have fever and neutropenia caused by a weakened immune system.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetics and serum levels of caspofungin acetate in immunocompromised children with new-onset fever and neutropenia.
* Determine the safety and tolerability of this drug in this patient population.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to age (2 to 11 vs 12 to 17).

Patients receive caspofungin acetate IV over 1 hour once daily for 4 to 28 days in the absence of the need to start standard empirical antifungal therapy, a breakthrough fungal infection, any deterioration of patient condition, or unacceptable toxicity.

Cohorts of 16 patients (8 per stratum) receive caspofungin acetate at 1 of 2 dose levels. Caspofungin acetate is escalated to dose level 2 if no more than 1 of 8 patients experiences dose-limiting toxicity at dose level 1.

Patients are followed at 14 days.

PROJECTED ACCRUAL: A total of 32-64 patients (16 per dose level (cohort), 8 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Immunocompromised with one or more of the following conditions:

  * Leukemia, lymphoma, or other cancer
  * Underwent bone marrow or peripheral blood stem cell transplantation
  * Aplastic anemia
* Planned chemotherapy likely to incur more than 10 days of neutropenia
* Absolute neutrophil count no greater than 500/mm^3 AND at least 1 recorded fever over 38.0 ° C within 24 hours of study
* No proven invasive fungal infection at time of study entry

  * Superficial fungal infection (e.g., cutaneous fungal infection, thrush, or candidal vaginitis) treatable with topical antifungals allowed

PATIENT CHARACTERISTICS:

Age:

* 2 to 17

Performance status:

* Not specified

Life expectancy:

* At least 5 days

Hematopoietic:

* See Disease Characteristics
* Hemodynamically stable with no hemodynamic compromise

Hepatic:

* AST or ALT no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN (unless related to bony metastases or other suspected bony processes)
* INR no greater than 1.6 (4.0 if receiving anticoagulants)
* No acute hepatitis or cirrhosis

Renal:

* Not specified

Other:

* Functioning central venous catheter in place
* No other condition or concurrent illness that would preclude study
* No prior allergy, hypersensitivity, or serious reaction to echinocandin antifungals
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception other than or in addition to oral contraceptives

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior enrollment into this study
* No more than 48 hours since prior parenteral systemic antibacterial therapy for fever and neutropenia
* At least 14 days since prior investigational antibiotic or antifungal drugs
* Concurrent topical antifungals (i.e., nystatin and/or azole formulations) for a superficial fungal infection allowed
* No other concurrent investigational drugs, including antibiotics or antifungals
* No concurrent rifampin, cyclosporine, phenytoin, carbamazapine, phenobarbital, or other antifungal treatments (except fluconazole)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2001-03; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Walsh, MD, Study Chair — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - St. Jude Children's Research Hospital, Memphis, Tennessee